CLINICAL TRIAL: NCT01966237
Title: USE OF ACUTE KIDNEY INJURY BIOMARKERS TO PREDICT IMPAIRED MILRINONE PHARMACOKINETICS IN CHILDREN FOLLOWING CARDIAC SURGERY
Brief Title: Milrinone Pharmacokinetics and Acute Kidney Injury
Acronym: MIL-PK
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-2507
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Congenital Heart Disease; Acute Kidney Injury
MeSH Terms: conditions — Heart Defects, Congenital; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute kidney injury: AKI defined by an elevation in urinary AKI biomarkers
- No acute kidney injury: No AKI defined by normal urinary AKI biomarkers

SUMMARY:
Acute kidney injury (AKI) occurs in 40% of children following heart surgery. Serum creatinine (Scr) is a late biomarker of AKI, rising 24-48 hours after surgery. Thus, for medicines excreted in the urine, AKI could potentially lead to toxic levels in the blood. Urinary biomarkers have the ability to detect AKI earlier. Whether early detection of AKI through urinary biomarkers can predict altered drug levels is unknown.

Milrinone is used to improve heart function after surgery, but accumulates in AKI resulting in low blood pressure. Dose adjustments are not currently possible because of the late rise in SCr, and are based on clinical parameters that may lead to clinically relevant over or under-dosing. Thus, this study will address an important knowledge gap being the first to use elevations of AKI biomarker concentrations to anticipate increased milrinone levels.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiothoracic surgery with cardiopulmonary bypass
* weight greater than 2500 grams (5 pounds 8 ounces) at the time of surgery
* gestational age > 36 weeks
* age less < to 1 year
* infants with complex congenital heart disease
* use of milrinone in the intra-operative and post-operative period.

Exclusion Criteria:

* Pre-existing kidney disease (structural and functional abnormalities) as determined by the Principal Investigator
* use of aminoglycosides within 48 hours of planned surgery
* cardiac arrest prior to cardiac surgery
* extracorporeal membrane oxygenation prior to cardiac surgery
* urinary tract infection prior to surgery
* repair of an isolated atrial or ventricular septal defect

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients less than or equal to 1 year who present for cardiac surgery at Cincinnati Children's Hospital Medical Center who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2013-09; Primary Completion 2017-07-31 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Biomarker elevation and milrinone clearance | By 24 hours
  The primary outcome variables for Aim 1 are an elevation in urinary AKI biomarkers to predict a 25% reduction in milrinone clearance.

SECONDARY OUTCOMES:
Creatinine elevation and milrinone clearance | by 72 hours
  The secondary outcome variables for Aim 2 include a 50-75% increase in SCr to predict a 25% reduction in milrinone clearance

OTHER OUTCOMES:
Hemodynamic parameters and AKI | by 72 hours
  Parameters of hemodynamic function defined by a decrease in central venous pressure of > 5cmH20, and/or a decrease in superior vena cava saturation by >10% at 12-36 hours after cardiopulmonary bypass. These surrogate markers of clinical outcome will be correlated with the following: operative mortality, longer time to achieve negative fluid balance, higher vasoactive inotrope score and longer intensive care and hospital length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Katja M Gist, DO, MSCS, Principal Investigator — University of Colorado, Denver
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Mizuno T, Gist KM, Gao Z, Wempe MF, Alten J, Cooper DS, Goldstein SL, Vinks AA. Developmental Pharmacokinetics and Age-Appropriate Dosing Design of Milrinone in Neonates and Infants with Acute Kidney Injury Following Cardiac Surgery. Clin Pharmacokinet. 2019 Jun;58(6):793-803. doi: 10.1007/s40262-018-0729-3. PMID 30607889
- [Derived] Gist KM, Cooper DS, Wrona J, Faubel S, Altmann C, Gao Z, Marino BS, Alten J, Hock KM, Mizuno T, Vinks AA, Joy MS, Wempe MF, Bennett MR, Goldstein SL. Acute Kidney Injury Biomarkers Predict an Increase in Serum Milrinone Concentration Earlier Than Serum Creatinine-Defined Acute Kidney Injury in Infants After Cardiac Surgery. Ther Drug Monit. 2018 Apr;40(2):186-194. doi: 10.1097/FTD.0000000000000496. PMID 29529007
- [Derived] Gist KM, Goldstein SL, Wrona J, Alten JA, Basu RK, Cooper DS, Soranno DE, Duplantis J, Altmann C, Gao Z, Faubel S. Kinetics of the cell cycle arrest biomarkers (TIMP-2*IGFBP-7) for prediction of acute kidney injury in infants after cardiac surgery. Pediatr Nephrol. 2017 Sep;32(9):1611-1619. doi: 10.1007/s00467-017-3655-y. Epub 2017 Apr 5. PMID 28382566